CLINICAL TRIAL: NCT05573958
Title: Open-label Randomized Control Trial to Assess the Efficacy and Safety of Dual Anticoagulants i.e. Rivaroxaban Plus Aspirin and Clopidogrel Plus Aspirin in Patients Suffering From an Acute Coronary Syndrome
Brief Title: To Assess the Efficacy and Safety of Dual Anticoagulants i.e. Rivaroxaban Plus Aspirin and Clopidogrel Plus Aspirin in Patients Suffering From an Acute Coronary Syndrome
Acronym: ACCP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sarmad Zahoor (Other)
Collaborators: University of Managemant and Technology, Pakistan (Unknown); Mayo Hospital Lahore (Other)
Responsible Party: Sponsor-Investigator, Sarmad Zahoor, Resident, Punjab Institute of Cardology
Organization: Punjab Institute of Cardology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIC-2022-06
Record Dates: First submitted 2022-09-09; First posted 2022-10-10 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Rivaroxaban; Clopidogrel; Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Rivaroxaban, Clopidogrel, and Aspirin (Experimental): Rivaroxaban 2.5 mg tablet twice daily orally, Clopidogrel 75 mg tablet once daily orally, and Aspirin 81 mg tablet once daily
  Interventions: Drug: Rivaroxaban 2.5 Mg Oral Tablet; Drug: Clopidogrel tablet; Drug: Aspirin tablet
- Arm B: Clopidogrel and Aspirin (Active Comparator): Clopidogrel 75 mg tablet once daily, and Aspirin 81 mg tablet once daily
  Interventions: Drug: Clopidogrel tablet; Drug: Aspirin tablet

INTERVENTIONS:
Drug: Rivaroxaban 2.5 Mg Oral Tablet — Rivaroxaban 2.5 mg oral tablet will be administered twice daily
  Other Names: Xarelto
  Arms: Arm A: Rivaroxaban, Clopidogrel, and Aspirin
Drug: Clopidogrel tablet — Clopidogrel 75 mg once daily orally
  Other Names: Plavix
Drug: Aspirin tablet — Aspirin 81 mg tablet once daily
  Other Names: Acetylsalicylic acid

SUMMARY:
Direct-acting oral anticoagulants (DOACs) have provided benefits to patients requiring anticoagulation for certain diseases by decreasing the burden of subcutaneous injections and the requirement for frequent monitoring through regular blood tests. DOACs do not require monitoring, have a more predictable pharmacokinetic (dosing) profile and have fewer interactions with other drugs. Various studies have reported the efficacy and safety of different dual-acting anticoagulants around the globe. However, there is little data available from Pakistan. Therefore, investigators propose this study to assess the efficiency and safety of rivaroxaban and clopidogrel along with aspirin in patients suffering from acute coronary syndrome. The objective of this study is to investigate the efficacy of dual anticoagulants i.e. aspirin plus rivaroxaban versus aspirin plus clopidogrel in patients suffering from acute coronary syndrome in terms of secondary prophylaxis. All the patient records will be documented in Case Report Form (CRF) at each visit. All data will be recorded in individual source documents. All CRF information is to be filled in by site staff. If an item is not available or is not applicable, this fact should be indicated. Blank spaces should not be present unless otherwise directed. The study monitor will perform source data verification of data entered into the CRF. The data entered into the CRF will be subject to data validation checks for consistency and completeness by the data management group. All CRFs should be maintained on the system with details of any changes logged accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged ≥ 18 years and above
* Participants able to understand the study procedures and willing to give written informed consent/assent to participate in the trial
* Participants willing to follow the study procedures of the study and available for the entire duration of the study.
* Female participants of childbearing potential must have a negative urine pregnancy test
* Women of childbearing potential (WOCBP) must be willing to abstain from heterosexual activities or agree to use highly effective, double-barrier contraception during the study and for 90 days following the final dose of study treatment, to avoid pregnancy. (This is in line with regulatory Guidance on Nonclinical Safety Studies for the Conduct of Human Clinical Trials and Marketing Authorization for Pharmaceuticals)

Exclusion Criteria:

* Co-morbidities: any pre-existing cardiac disease, pulmonary disease, diabetes
* Arrhythmias
* Pre-existing hepatic disease
* Pre-existing renal disease
* Already taking any drug
* Pregnancy
* Thyroid dysfunctions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 3 months
  Myocardial infarction, Arrhythmia, Stroke, Pulmonary Edema, Death

IPD SHARING:
Plan to Share IPD: No